CLINICAL TRIAL: NCT05825001
Title: Pilot Study of Episodic Future Thinking Among Cigarette Smokers
Brief Title: Evaluating the Episodic Future Thinking Intervention for Reducing Cigarette Consumption in Cigarette Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 2684022
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (active EFT) (Experimental): Participants receive the active EFT stimulus and use the iCOquit Smokerlyzer carbon monoxide monitor on study.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Medical Device Usage and Evaluation
- Arm II (control EFT) (Active Comparator): Participants receive the control EFT stimulus and use the iCOquit Smokerlyzer carbon monoxide monitor on study.
  Interventions: Behavioral: Smoking Cessation Intervention (control); Other: Medical Device Usage and Evaluation

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention — Receive active EFT stimulus
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm 1 (active EFT)
Behavioral: Smoking Cessation Intervention (control) — Receive control EFT stimulus
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm II (control EFT)
Other: Medical Device Usage and Evaluation — Use iCOquit Smokerlyzer carbon monoxide monitor

SUMMARY:
This clinical trial evaluates the effectiveness of active episodic future thinking (EFT) stimuli for reducing cigarette consumption in cigarette smokers. EFT is an innovative framing method shown to significantly activate brain regions involved in future thinking, planning, and other executive functions. Active EFT stimuli are positive events, unrelated to smoking, that participants anticipate, look forward to, and can vividly imagine happening up to 1 year in the future. Control EFT stimuli are positive past events, unrelated to smoking, that participants can vividly remember happening in the recent past. Active EFT stimuli may help reduce cigarette consumption among cigarette smokers by exposing them to personally relevant future oriented stimuli.

DETAILED DESCRIPTION:
PRIMARY OBJEECTIVE:

I. To evaluate the efficacy of episodic future thinking (EFT) for smoking cessation.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (ACTIVE): Participants receive the active EFT stimulus and use the iCOquit Smokerlyzer carbon monoxide monitor on study.

ARM II (CONTROL): Participants receive the control EFT stimulus and use the iCOquit Smokerlyzer carbon monoxide monitor on study.

ELIGIBILITY:
Inclusion Criteria:

* Smoke >= 10 cigarettes daily
* >32 on the Vividness of Visual Imagery Questionnaire (VVIQ)
* No regular use of other tobacco products
* In possession of a smartphone with text messaging capabilities

  * Willing to quit smoking in the next 30 days
  * Low socioeconomic status
  * Veteran of the US armed services

Exclusion Criteria:

* Unable or unwilling to provide verbal consent
* Unable or unwilling to provide data to the research team
* Current use of nicotine replacement therapy, bupropion, or varenicline
* Use of drugs of abuse in the past 30 days
* Living in the same household as a participant already enrolled in this study
* Unable or unwilling to use nicotine patches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of carbon monoxide on breath | From baseline up to 30 days
  Will be measured by Micro+Basic carbon monoxide monitor

SECONDARY OUTCOMES:
Reduction in delay discounting rate | Up to 30 days
  participants will be guided to imagine the situational and sensory details for each of the stimuli until the vividness scores are ≥ 4 on a scale of 1-5 (1=very low, 5=very high).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sheffer, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided